CLINICAL TRIAL: NCT00141973
Title: Time Course of Procalcitonin and C Reactive Protein in Septic Patients Under Treatment With Corticosteroids
Status: Completed | Type: Observational
Sponsor: Ospedale Regionale Bellinzona e Valli (Other)
Collaborators: Brahms SA, D-16761 Hennigsdorf bei Berlin (Unknown)
Other Study IDs: CE1408
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2008-05-14 (Estimated); Status verified 2008-05

CONDITIONS: Sepsis
Keywords: Procalcitonin; Sepsis; Corticosteroids
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
A systemic treatment with corticosteroids has been advocated for various bacterial infectious diseases. Since the production of CRP is down-regulated by corticosteroids, a smaller increase or a more rapid decrease of this acute phase protein will:

1. suggest attenuated systemic inflammation, but
2. does not necessarily reflect adequate therapy of the infection.

For several reasons (good diagnostic tool for sepsis, induction not decreased by immunosuppressive therapy), procalcitonin could be a better marker for activity of sepsis in patients under corticosteroids. As this issue has not yet been examined the investigators will prospectively study the time-course of PTC and CRP in a well-defined septic patient group, that in adjunction to antibiotic therapy also received systemic corticosteroid treatment and compare it to a similar group without corticosteroid treatment.

ELIGIBILITY:
Inclusion Criteria:

* Acute exacerbation of chronic obstructive pulmonary disease (COPD) due to bacterial pneumonia

Exclusion Criteria:

* Chronic systemic use of corticosteroids

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-11; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Perren, MD, Principal Investigator — Ospedale Regionale Bellinzona e Valli, CH-6500 Bellinzona
Locations (1):
- Ospedale Regionale Bellinzona e Valli, Bellinzona, Canton Ticino, Switzerland